CLINICAL TRIAL: NCT04718870
Title: Open-label Exploratory Study to Evaluate the Effect of Dupilumab on Skin Barrier Function in Pediatric Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Dupilumab-PEdiatric Skin Barrier Function and LIpidomics STudy in Patients With Atopic Dermatitis
Acronym: PELISTAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS16764; 2020-001518-40 (EudraCT Number); U1111-1255-4378 (Other: UTN)
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Results first posted 2023-10-17 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Dermatitis Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Atopic Dermatitis Participants (Experimental): Pediatric participants with moderate-to-severe atopic dermatitis (AD) and with baseline body weight more than or equal to (>=) 15 kilograms (kg) and less than (<) 30 kg received a subcutaneous (SC) loading dose of dupilumab 600 milligrams (mg) (2 injections of dupilumab 300 mg) on Day 1 (Week 0) followed by dupilumab 300 mg SC injection every 4 weeks (Q4W), from Week 4 to Week 12. Pediatric participants with body weight >=30 kg and <60 kg received SC loading dose of dupilumab 400 mg (2 injections of dupilumab 200 mg) on Day 1 (Week 0), followed by dupilumab 200 mg SC injection every 2 weeks (Q2W), from Week 2 to Week 14.
  Interventions: Drug: Dupilumab SAR231893
- Healthy Volunteers (No Intervention): Healthy volunteers with age, gender, location of targeted skin lesion area and study site matched to selected AD participants, received no treatment, but were monitored in a similar way as AD participants.

INTERVENTIONS:
Drug: Dupilumab SAR231893 — Pharmaceutical form: solution for injection Route of administration: subcutaneous (SC)
  Other Names: REGN668
  Arms: Atopic Dermatitis Participants

SUMMARY:
Primary Objective:

- Evaluate changes in skin barrier function with transepidermal water loss (TEWL) assessed after skin tape stripping (STS) in predefined lesional skin in pediatric participants with moderate to severe atopic dermatitis (AD) treated with dupilumab.

Secondary Objectives:

* Evaluate changes in skin barrier function with TEWL assessed after STS in predefined lesional and non-lesional skin in pediatric participants with moderate to severe AD treated with dupilumab in reference to normal skin of healthy volunteers.
* Evaluate time course of change in skin barrier function with TEWL assessed before and after STS in predefined lesional and non-lesional skin in pediatric participants with moderate to severe AD during dupilumab treatment phase and follow-up period in reference to normal skin of healthy volunteers.

DETAILED DESCRIPTION:
Total study duration including screening and follow-up was 32 weeks.

ELIGIBILITY:
Inclusion criteria :

* Participant must be between >=6 to <12 years of age (inclusive), at the time of signing the informed consent
* 15 kg <= body weight <60 kg.

Atopic dermatitis participants:

* Male or female pediatric participants.
* Participants with AD diagnosis according to Hanifin and Rajka criteria at least 1 year before screening.
* Investigator Global Assessment (IGA) score of >=3 (for US participants) or IGA >=4 (for EU participants) at screening (on the 0-4 scale) depending on approved label indication in the country.
* Participants with moderate to severe AD those were eligible to be treated with dupilumab according to product label.
* Participants with AD must have had active lesions on the upper limbs or lower limbs (including trunk, if needed), with severity for lesion erythema or edema/papulation >=2 at screening on the 0-3 scale of the Individual Signs Score.
* Participants should have had a non-lesional (normal looking) skin area 4 centimeter (cm) from the edge of the lesional area. If unable to identify non-lesional skin 4 cm from the lesional area, it was acceptable to identify normal looking skin as close to the lesion as possible.

Healthy volunteers:

- Age and gender matched (match on age ±2 years) to a selected AD participant by study site.

Exclusion criteria:

* Previous treatment with dupilumab within 6 months prior to screening.
* Skin conditions other than AD that can confound assessments in the area of TEWL assessments in the opinion of the Investigator (i.e., skin atrophy, ichthyosis, tinea infection, contact dermatitis).
* Cracked, crusted, oozing, or bleeding AD lesions in the designated lesional assessment area leaving insufficient skin that was adequate for TEWL assessments.
* Hypersensitivity to the active substance or to any of the excipients of dupilumab.
* Ocular disorder that in the opinion of the Investigator could adversely affect the individual's risk for study participation. Examples include -but are not limited to- individuals with a history of active cases of herpes keratitis; Sjogren's syndrome, keratoconjunctivitis sicca, or individuals with ocular conditions that require the use of ocular corticosteroids or cyclosporine.
* Healthy volunteers with a personal history of an atopic condition.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- United States (2):
  - Investigational Site Number :8400002, Los Angeles, California
  - Investigational Site Number :8400001, Denver, Colorado
- Investigational Site Number :8260001, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS16764 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25291&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 3 active sites in the United States and United Kingdom. A total of 43 participants were screened between 19 Feb 2021 and 12 May 2022, out of which 41 were enrolled and 2 were screen failures due to not meeting inclusion criteria.
Pre-assignment Details: Healthy volunteer's cohort received no treatment and was considered as a reference comparator group.
Groups:
- Healthy Volunteers: Healthy volunteers with age, gender, location of targeted skin lesion area and study site matched to selected atopic dermatitis (AD) participants, received no treatment, but were monitored in a similar way as AD participants.
- Atopic Dermatitis Participants: Pediatric participants with moderate-to-severe AD and with baseline body weight more than or equal to (>=) 15 kilograms (kg) and less than (<) 30 kg received a subcutaneous (SC) loading dose of dupilumab 600 milligrams (mg) (2 injections of dupilumab 300 mg) on Day 1 (Week 0) followed by dupilumab 300 mg SC injection every 4 weeks (Q4W), from Week 4 to Week 12. Pediatric participants with body weight >=30 kg and <60 kg received SC loading dose of dupilumab 400 mg (2 injections of dupilumab 200 mg) on Day 1 (Week 0), followed by dupilumab 200 mg SC injection every 2 weeks (Q2W), from Week 2 to Week 14.
Period: Overall Study
Arm/Group | Healthy Volunteers | Atopic Dermatitis Participants
Started | 18 | 23
Completed | 18 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on modified intent-to-treat (mITT) population which included all enrolled AD participants who received at least 1 dose of investigational medicinal product (IMP) and all enrolled healthy volunteers who had at least 1 TEWL/STS assessment performed, irrespective of compliance with protocol and procedures. If prohibited therapies used for AD, only visits prior to rescue treatment were considered.
Groups:
- Atopic Dermatitis Participants: Pediatric participants with moderate-to-severe AD and with baseline body weight >=15 kg and <30 kg received a SC loading dose of dupilumab 600 mg (2 injections of dupilumab 300 mg) on Day 1 (Week 0) followed by dupilumab 300 mg SC injection Q4W, from Week 4 to Week 12. Pediatric participants with body weight >=30 kg and <60 kg received SC loading dose of dupilumab 400 mg (2 injections of dupilumab 200 mg) on Day 1 (Week 0), followed by dupilumab 200 mg SC injection Q2W, from Week 2 to Week 14.
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Atopic Dermatitis Participants | Total
Number analyzed (Participants) | 18 | 23 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.2 (1.8) | 7.8 (1.6) | 8.0 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 10 | 15 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 9 | 16 | 25
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Transepidermal Water Loss (TEWL) After 5 Skin Tape Stripping (STS) on Lesional Skin (LS) in AD Participants at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize skin barrier function (SBF). TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. Lesional skin (LS) areas for TEWL assessment and STS was identified at Baseline ('predefined skin area'). Within the predefined LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on the first spot. Percent Change from Baseline at Week 16 in TEWL after 5 STS on LS (first spot) in AD participants were reported in this outcome measure (OM).
Time Frame: Baseline, Week 16
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' = participants with available data for this OM. Data for this OM was not planned to be collected and analyzed for Healthy Volunteer arm as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 18
percent change | -38.5633 (27.1211)

2. Secondary Outcome: Percent Change From Baseline in TEWL After 20 STS on Lesional Skin in AD Participants at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The LS areas for TEWL assessment and STS were identified at Baseline (predefined skin area). Within the predefined LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS areas at specified time points. STS assessment at baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent change from baseline at Week 16 in TEWL after 20 STS on LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' = participants with available data for this OM. Data for this OM was not planned to be collected and analyzed for healthy volunteer arm as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 17
percent change | -33.1336 (28.1613)

3. Secondary Outcome: Absolute Change From Baseline in TEWL After 20 STS on Lesional Skin in AD Participants at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that was used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The LS areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS areas at specified time points. STS assessment at baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Absolute change from Baseline at Week 16 in TEWL after 20 STS on LS (first spot) in AD participants were reported in this OM
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 17
grams per square meter per hour | -35.6671 (31.2267)

4. Secondary Outcome: Percent Change From Baseline in TEWL After 20 STS on Non-lesional Skin (Non-LS) in AD Participants at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The non-LS areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined non-LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined non-LS areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent change from Baseline at Week 16 in TEWL after 20 STS on non-LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 17
percent change | -6.1452 (67.9496)

5. Secondary Outcome: Absolute Change From Baseline in TEWL After 20 STS on Non-lesional Skin in AD Participants at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The non-LS areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined non-LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined non-LS areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on the first spot. Absolute change from baseline at Week 16 in TEWL after 20 STS on non-LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 17
grams per square meter per hour | -13.6682 (33.3065)

6. Secondary Outcome: Percent Change From Baseline in TEWL After 20 STS on Normal Skin in Healthy Volunteers at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The normal skin areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined normal skin areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent change from baseline at Week 16 in TEWL after 20 STS on normal skin (first spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Week 16
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' = participants with available data for this OM. Data for this OM was not planned to be collected and analyzed for atopic dermatitis participant arm as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 11
percent change | 13.2578 (64.3880)

7. Secondary Outcome: Absolute Change From Baseline in TEWL After 20 STS on Normal Skin in Healthy Volunteers at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The normal skin areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined normal skin areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Absolute change from baseline at Week 16 in TEWL after 20 STS on normal skin (first spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 11
grams per square meter per hour | 5.9327 (32.0123)

8. Secondary Outcome: Percent Change From Baseline in TEWL After 15 STS on Lesional Skin in AD Participants at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The LS areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS and non-LS areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent change from baseline at Week 16 in TEWL after 15 STS on LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 18
percent change | -33.3119 (32.7125)

9. Secondary Outcome: Absolute Change From Baseline in TEWL After 15 STS on Lesional Skin in AD Participants at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The LS areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS areas at specified time points. STS assessment at Baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Absolute change from baseline at Week 16 in TEWL after 15 STS on LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 18
grams per square meter per hour | -33.4028 (31.1957)

10. Secondary Outcome: Percent Change From Baseline in TEWL After 15 STS on Non-lesional Skin in AD Participants at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The non-LS areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined non-LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined non-LS areas at specified time points. STS assessment at baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent change from baseline at Week 16 in TEWL after 15 STS on non-LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 17
percent change | -7.6067 (54.7945)

11. Secondary Outcome: Absolute Change From Baseline in TEWL After 15 STS on Non-lesional Skin in AD Participants at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The non-LS areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined non-LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined non-LS areas at specified time points. STS assessment at baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Absolute change from baseline at Week 16 in TEWL after 15 STS on non-LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' = participants with available data for this OM. Data for this OM was not planned to be collected and analyzed for 'healthy volunteer' arm as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 17
grams per square meter per hour | -12.6576 (30.0412)

12. Secondary Outcome: Percent Change From Baseline in TEWL After 15 STS on Normal Skin in Healthy Volunteers at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The normal skin areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined normal skin areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment at baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent change from baseline at Week 16 in TEWL after 15 STS on normal skin (first spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Week 16
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' = participants with available data for this OM. Data for this OM was not planned to be collected and analyzed for atopic dermatitis participants arm as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 11
percent change | 4.5364 (42.7525)

13. Secondary Outcome: Absolute Change From Baseline in TEWL After 15 STS on Normal Skin in Healthy Volunteers at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The normal skin areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined normal skin areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment at baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Absolute change from baseline at Week 16 in TEWL after 15 STS on normal skin (first spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 11
grams per square meter per hour | 0.1082 (17.5865)

14. Secondary Outcome: Percent Change From Baseline in TEWL After 10 STS on Lesional Skin in AD Participants at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The LS areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS areas at specified time points. STS assessment at baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent change from baseline at Week 16 in TEWL after 10 STS on LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 17
percent change | -34.7741 (31.0541)

15. Secondary Outcome: Absolute Change From Baseline in TEWL After 10 STS on Lesional Skin in AD Participants at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The LS areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS areas at specified time points. STS assessment at baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Absolute change from baseline at Week 16 in TEWL after 10 STS on LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 17
grams per square meter per hour | -33.1024 (36.2286)

16. Secondary Outcome: Percent Change From Baseline in TEWL After 10 STS on Non-lesional Skin in AD Participants at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The non-LS areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined non-LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined non-LS areas at specified time points. STS assessment at baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent change from baseline at Week 16 in TEWL after 10 STS on non-LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 17
percent change | -3.8193 (74.6263)

17. Secondary Outcome: Absolute Change From Baseline in TEWL After 10 STS on Non-lesional Skin in AD Participants at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The non-LS areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined non-LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined non-LS areas at specified time points. STS assessment at baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Absolute change from baseline at Week 16 in TEWL after 10 STS on non-LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 17
grams per square meter per hour | -10.9488 (31.1300)

18. Secondary Outcome: Percent Change From Baseline in TEWL After 10 STS on Normal Skin in Healthy Volunteers at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The normal skin areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined normal skin areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment at baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent change from baseline at Week 16 in TEWL after 10 STS on normal skin (first spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 11
percent change | 0.7091 (25.0615)

19. Secondary Outcome: Absolute Change From Baseline in TEWL After 10 STS on Normal Skin in Healthy Volunteers at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The normal skin areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined normal skin areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment at baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Absolute change from baseline at Week 16 in TEWL after 10 STS on normal skin (first spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 11
grams per square meter per hour | -1.3482 (6.6778)

20. Secondary Outcome: Percent Change From Baseline in TEWL After 5 STS on Non-lesional Skin in AD Participants at Week16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The non-LS areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined non-LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined non-LS areas at specified time points. STS assessment at baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent change from baseline at Week 16 in TEWL after 5 STS on non-LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 17
percent change | -4.8842 (70.5670)

21. Secondary Outcome: Absolute Change From Baseline in TEWL After 5 STS on Non-lesional Skin in AD Participants at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The non-LS areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined non-LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined non-LS areas at specified time points. STS assessment at baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Absolute change from baseline at Week 16 in TEWL after 5 STS on non-LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 17
grams per square meter per hour | -9.0771 (21.3022)

22. Secondary Outcome: Percent Change From Baseline in TEWL After 5 STS on Normal Skin in Healthy Volunteers at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The normal skin areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined normal skin areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment at baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Percent change from baseline at Week 16 in TEWL after 5 STS on normal skin (first spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Week 16
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' = participants with available data for this OM. Data for this OM was not planned to be collected and analyzed for atopic dermatitis arm as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 11
percent change | 1.4464 (26.7257)

23. Secondary Outcome: Absolute Change From Baseline in TEWL After 5 STS on Normal Skin in Healthy Volunteers at Week 16
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of the skin are peeled away using adhesive discs. The normal skin areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined normal skin areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment at baseline (Week 0, Day 1) and Week 16 was conducted on first spot. Absolute change from baseline at Week 16 in TEWL after 5 STS on normal skin (first spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Week 16
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 11
grams per square meter per hour | -1.0255 (4.3657)

24. Secondary Outcome: Percent Change From Baseline in TEWL Before STS on Lesional Skin in AD Participants at Days 8, 15, 22, 29, 43, 57, 85, 113, 155 and 197
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. LS areas for TEWL assessment were identified at baseline ('predefined skin area'). Within predefined LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS on pre-defined LS areas at specified time points. At each visit, before STS, all three spots were assessed. Percent change from Baseline at specified time points in TEWL before STS on LS (at each spot) in AD participants were reported in this OM.
Time Frame: Baseline, Days 8, 15, 22, 29, 43, 57, 85, 113, 155 and 197
Population: Analysis was performed on mITT population. Here, 'number analyzed' = participants with available data for each specified category. Data for this OM was not planned to be collected and analyzed for 'healthy volunteer' arm as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 23
percent change
  Day 8 - Spot 1: number analyzed (Participants) | 22
  Day 8 - Spot 1 | -7.1596 (36.6637)
  Day 8 - Spot 2 | -6.3439 (33.8145)
  Day 8 - Spot 3 | -7.0747 (28.3554)
  Day 15 - Spot 1: number analyzed (Participants) | 22
  Day 15 - Spot 1 | -15.3096 (45.6163)
  Day 15 - Spot 2: number analyzed (Participants) | 22
  Day 15 - Spot 2 | -11.0740 (35.5483)
  Day 15 - Spot 3: number analyzed (Participants) | 22
  Day 15 - Spot 3 | -8.1780 (44.9382)
  Day 22 - Spot 1: number analyzed (Participants) | 21
  Day 22 - Spot 1 | -30.3070 (33.6643)
  Day 22 - Spot 2: number analyzed (Participants) | 21
  Day 22 - Spot 2 | -29.1730 (31.7167)
  Day 22 - Spot 3: number analyzed (Participants) | 21
  Day 22 - Spot 3 | -27.0015 (25.8528)
  Day 29 - Spot 1: number analyzed (Participants) | 20
  Day 29 - Spot 1 | -37.8349 (24.7709)
  Day 29 - Spot 2: number analyzed (Participants) | 20
  Day 29 - Spot 2 | -33.0139 (27.8560)
  Day 29 - Spot 3: number analyzed (Participants) | 20
  Day 29 - Spot 3 | -32.7080 (28.8445)
  Day 43 - Spot 1: number analyzed (Participants) | 17
  Day 43 - Spot 1 | -37.8675 (29.0275)
  Day 43 - Spot 2: number analyzed (Participants) | 17
  Day 43 - Spot 2 | -36.1625 (28.9829)
  Day 43 - Spot 3: number analyzed (Participants) | 17
  Day 43 - Spot 3 | -32.9996 (33.2028)
  Day 57 - Spot 1: number analyzed (Participants) | 19
  Day 57 - Spot 1 | -38.2449 (40.0558)
  Day 57 - Spot 2: number analyzed (Participants) | 19
  Day 57 - Spot 2 | -39.3104 (27.6888)
  Day 57 - Spot 3: number analyzed (Participants) | 19
  Day 57 - Spot 3 | -35.8992 (27.9526)
  Day 85 - Spot 1: number analyzed (Participants) | 18
  Day 85 - Spot 1 | -45.6060 (23.2839)
  Day 85 - Spot 2: number analyzed (Participants) | 18
  Day 85 - Spot 2 | -40.8609 (30.8002)
  Day 85 - Spot 3: number analyzed (Participants) | 18
  Day 85 - Spot 3 | -41.1371 (24.5842)
  Day 113 - Spot 1: number analyzed (Participants) | 18
  Day 113 - Spot 1 | -36.0863 (33.7259)
  Day 113 - Spot 2: number analyzed (Participants) | 18
  Day 113 - Spot 2 | -37.4815 (30.8507)
  Day 113 - Spot 3: number analyzed (Participants) | 18
  Day 113 - Spot 3 | -32.3491 (29.2966)
  Day 155 - Spot 1: number analyzed (Participants) | 14
  Day 155 - Spot 1 | -40.9536 (30.9966)
  Day 155 - Spot 2: number analyzed (Participants) | 14
  Day 155 - Spot 2 | -20.8463 (50.6518)
  Day 155 - Spot 3: number analyzed (Participants) | 14
  Day 155 - Spot 3 | -31.3185 (42.0614)
  Day 197 - Spot 1: number analyzed (Participants) | 15
  Day 197 - Spot 1 | -35.2305 (45.8818)
  Day 197 - Spot 2: number analyzed (Participants) | 15
  Day 197 - Spot 2 | -30.3358 (48.3028)
  Day 197 - Spot 3: number analyzed (Participants) | 15
  Day 197 - Spot 3 | -36.5267 (37.7230)

25. Secondary Outcome: Absolute Change From Baseline in TEWL Before STS on Lesional Skin in AD Participants at Days 8, 15, 22, 29, 43, 57, 85, 113, 155 and 197
Description: TEWL assessment: noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. LS areas for TEWL assessment were identified at baseline (predefined skin area). Within predefined LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS on pre-defined LS areas at specified time points. At each visit, before STS, all three spots were assessed. Absolute change from baseline at specified time points in TEWL before STS on LS (at each spot) in AD participants were reported in this OM.
Time Frame: Baseline, Days 8, 15, 22, 29, 43, 57, 85, 113, 155 and 197
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 23
grams per square meter per hour
  Day 8 - Spot 1: number analyzed (Participants) | 22
  Day 8 - Spot 1 | -9.3486 (21.2256)
  Day 8 - Spot 2 | -6.0491 (17.5810)
  Day 8 - Spot 3 | -3.1965 (14.4640)
  Day 15 - Spot 1: number analyzed (Participants) | 22
  Day 15 - Spot 1 | -15.4336 (25.0975)
  Day 15 - Spot 2: number analyzed (Participants) | 22
  Day 15 - Spot 2 | -9.8073 (19.7385)
  Day 15 - Spot 3: number analyzed (Participants) | 22
  Day 15 - Spot 3 | -7.6682 (21.9239)
  Day 22 - Spot 1: number analyzed (Participants) | 21
  Day 22 - Spot 1 | -23.0157 (26.8847)
  Day 22 - Spot 2: number analyzed (Participants) | 21
  Day 22 - Spot 2 | -20.7186 (23.4149)
  Day 22 - Spot 3: number analyzed (Participants) | 21
  Day 22 - Spot 3 | -15.6557 (20.1212)
  Day 29 - Spot 1: number analyzed (Participants) | 20
  Day 29 - Spot 1 | -23.9585 (21.7106)
  Day 29 - Spot 2: number analyzed (Participants) | 20
  Day 29 - Spot 2 | -21.2010 (21.2593)
  Day 29 - Spot 3: number analyzed (Participants) | 20
  Day 29 - Spot 3 | -17.9170 (19.7310)
  Day 43 - Spot 1: number analyzed (Participants) | 17
  Day 43 - Spot 1 | -27.0535 (28.0249)
  Day 43 - Spot 2: number analyzed (Participants) | 17
  Day 43 - Spot 2 | -24.5188 (25.6684)
  Day 43 - Spot 3: number analyzed (Participants) | 17
  Day 43 - Spot 3 | -20.7018 (22.5936)
  Day 57 - Spot 1: number analyzed (Participants) | 19
  Day 57 - Spot 1 | -25.1221 (27.0210)
  Day 57 - Spot 2: number analyzed (Participants) | 19
  Day 57 - Spot 2 | -24.2358 (24.6028)
  Day 57 - Spot 3: number analyzed (Participants) | 19
  Day 57 - Spot 3 | -20.3379 (20.3751)
  Day 85 - Spot 1: number analyzed (Participants) | 18
  Day 85 - Spot 1 | -29.1917 (24.3114)
  Day 85 - Spot 2: number analyzed (Participants) | 18
  Day 85 - Spot 2 | -24.4494 (24.2054)
  Day 85 - Spot 3: number analyzed (Participants) | 18
  Day 85 - Spot 3 | -23.1056 (20.4692)
  Day 113 - Spot 1: number analyzed (Participants) | 18
  Day 113 - Spot 1 | -24.6678 (27.8013)
  Day 113 - Spot 2: number analyzed (Participants) | 18
  Day 113 - Spot 2 | -23.2878 (26.5670)
  Day 113 - Spot 3: number analyzed (Participants) | 18
  Day 113 - Spot 3 | -17.9028 (22.2483)
  Day 155 - Spot 1: number analyzed (Participants) | 14
  Day 155 - Spot 1 | -28.2564 (29.2212)
  Day 155 - Spot 2: number analyzed (Participants) | 14
  Day 155 - Spot 2 | -18.7786 (31.4917)
  Day 155 - Spot 3: number analyzed (Participants) | 14
  Day 155 - Spot 3 | -19.8921 (27.8520)
  Day 197 - Spot 1: number analyzed (Participants) | 15
  Day 197 - Spot 1 | -27.4493 (33.7080)
  Day 197 - Spot 2: number analyzed (Participants) | 15
  Day 197 - Spot 2 | -22.5607 (31.7696)
  Day 197 - Spot 3: number analyzed (Participants) | 15
  Day 197 - Spot 3 | -22.0860 (27.1286)

26. Secondary Outcome: Percent Change From Baseline in TEWL Before STS on Non-lesional Skin in AD Participants at Days 8, 15, 22, 29, 43, 57, 85, 113, 155 and 197
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. Non-LS areas for TEWL assessment were identified at baseline (predefined skin area). Within predefined non-LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS on pre-defined non-LS areas at specified time points. At each visit, before STS, all three spots were assessed. Percent change from baseline at specified time points in TEWL before STS on non-LS (at each spot) in AD participants were reported in this OM.
Time Frame: Baseline, Days 8, 15, 22, 29, 43, 57, 85, 113, 155 and 197
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 23
percent change
  Day 8 - Spot 1 | 41.0825 (91.3744)
  Day 8 - Spot 2: number analyzed (Participants) | 21
  Day 8 - Spot 2 | 13.5236 (49.3733)
  Day 8 - Spot 3 | 9.7943 (43.9272)
  Day 15 - Spot 1: number analyzed (Participants) | 22
  Day 15 - Spot 1 | 19.0612 (58.1703)
  Day 15 - Spot 2: number analyzed (Participants) | 21
  Day 15 - Spot 2 | 9.6866 (52.6831)
  Day 15 - Spot 3: number analyzed (Participants) | 21
  Day 15 - Spot 3 | 13.2574 (55.8095)
  Day 22 - Spot 1: number analyzed (Participants) | 21
  Day 22 - Spot 1 | -3.9277 (35.9880)
  Day 22 - Spot 2: number analyzed (Participants) | 20
  Day 22 - Spot 2 | 8.9306 (70.2617)
  Day 22 - Spot 3: number analyzed (Participants) | 21
  Day 22 - Spot 3 | 0.4973 (49.5636)
  Day 29 - Spot 1: number analyzed (Participants) | 20
  Day 29 - Spot 1 | -8.9585 (39.0443)
  Day 29 - Spot 2: number analyzed (Participants) | 19
  Day 29 - Spot 2 | -10.5728 (35.2672)
  Day 29 - Spot 3: number analyzed (Participants) | 20
  Day 29 - Spot 3 | -13.0407 (44.5264)
  Day 43 - Spot 1: number analyzed (Participants) | 17
  Day 43 - Spot 1 | -15.6919 (29.7995)
  Day 43 - Spot 2: number analyzed (Participants) | 16
  Day 43 - Spot 2 | -21.6885 (30.1255)
  Day 43 - Spot 3: number analyzed (Participants) | 17
  Day 43 - Spot 3 | -16.2025 (42.7984)
  Day 57 - Spot 1: number analyzed (Participants) | 19
  Day 57 - Spot 1 | -24.5008 (26.9801)
  Day 57 - Spot 2: number analyzed (Participants) | 18
  Day 57 - Spot 2 | -27.6040 (23.0969)
  Day 57 - Spot 3: number analyzed (Participants) | 19
  Day 57 - Spot 3 | -25.7321 (33.1310)
  Day 85 - Spot 1: number analyzed (Participants) | 18
  Day 85 - Spot 1 | -21.9316 (34.3620)
  Day 85 - Spot 2: number analyzed (Participants) | 17
  Day 85 - Spot 2 | -16.7008 (62.4384)
  Day 85 - Spot 3: number analyzed (Participants) | 18
  Day 85 - Spot 3 | -29.2721 (40.0673)
  Day 113 - Spot 1: number analyzed (Participants) | 17
  Day 113 - Spot 1 | -20.4359 (42.6948)
  Day 113 - Spot 2: number analyzed (Participants) | 16
  Day 113 - Spot 2 | -23.1303 (41.2717)
  Day 113 - Spot 3: number analyzed (Participants) | 17
  Day 113 - Spot 3 | -27.4981 (33.5326)
  Day 155 - Spot 1: number analyzed (Participants) | 14
  Day 155 - Spot 1 | -6.7535 (73.4261)
  Day 155 - Spot 2: number analyzed (Participants) | 13
  Day 155 - Spot 2 | -16.3903 (41.9864)
  Day 155 - Spot 3: number analyzed (Participants) | 14
  Day 155 - Spot 3 | -19.3970 (46.5302)
  Day 197 - Spot 1: number analyzed (Participants) | 16
  Day 197 - Spot 1 | -23.3812 (39.5978)
  Day 197 - Spot 2: number analyzed (Participants) | 15
  Day 197 - Spot 2 | -27.3104 (32.8267)
  Day 197 - Spot 3: number analyzed (Participants) | 16
  Day 197 - Spot 3 | -22.1813 (40.5124)

27. Secondary Outcome: Absolute Change From Baseline in TEWL Before STS on Non-lesional Skin in AD Participants at Days 8, 15, 22, 29, 43, 57, 85, 113, 155 and 197
Description: TEWL assessment: noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. Non-LS areas for TEWL assessment were identified at baseline (predefined skin area). Within predefined non-LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS on pre-defined non-LS areas at specified time points. At each visit, before STS, all three spots were assessed. Absolute change from baseline at specified time points in TEWL before STS on non-LS (at each spot) in AD participants were reported in this OM.
Time Frame: Baseline, Days 8, 15, 22, 29, 43, 57, 85, 113, 155 and 197
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 23
grams per square meter per hour
  Day 8 - Spot 1 | 4.1752 (14.1047)
  Day 8 - Spot 2: number analyzed (Participants) | 21
  Day 8 - Spot 2 | -0.0248 (11.8585)
  Day 8 - Spot 3 | -0.3413 (9.8571)
  Day 15 - Spot 1: number analyzed (Participants) | 22
  Day 15 - Spot 1 | 0.4723 (9.7975)
  Day 15 - Spot 2: number analyzed (Participants) | 21
  Day 15 - Spot 2 | -2.6176 (13.1001)
  Day 15 - Spot 3: number analyzed (Participants) | 21
  Day 15 - Spot 3 | -1.0171 (11.3877)
  Day 22 - Spot 1: number analyzed (Participants) | 21
  Day 22 - Spot 1 | -3.8162 (10.3046)
  Day 22 - Spot 2: number analyzed (Participants) | 20
  Day 22 - Spot 2 | -3.5735 (16.4593)
  Day 22 - Spot 3: number analyzed (Participants) | 21
  Day 22 - Spot 3 | -5.3314 (12.8392)
  Day 29 - Spot 1: number analyzed (Participants) | 20
  Day 29 - Spot 1 | -5.3400 (10.8674)
  Day 29 - Spot 2: number analyzed (Participants) | 19
  Day 29 - Spot 2 | -6.7411 (13.5999)
  Day 29 - Spot 3: number analyzed (Participants) | 20
  Day 29 - Spot 3 | -9.5905 (14.0754)
  Day 43 - Spot 1: number analyzed (Participants) | 17
  Day 43 - Spot 1 | -6.7424 (9.7834)
  Day 43 - Spot 2: number analyzed (Participants) | 16
  Day 43 - Spot 2 | -8.8444 (12.4876)
  Day 43 - Spot 3: number analyzed (Participants) | 17
  Day 43 - Spot 3 | -10.5600 (14.1984)
  Day 57 - Spot 1: number analyzed (Participants) | 19
  Day 57 - Spot 1 | -8.2874 (8.5546)
  Day 57 - Spot 2: number analyzed (Participants) | 18
  Day 57 - Spot 2 | -9.7772 (11.7879)
  Day 57 - Spot 3: number analyzed (Participants) | 19
  Day 57 - Spot 3 | -11.9179 (13.1662)
  Day 85 - Spot 1: number analyzed (Participants) | 18
  Day 85 - Spot 1 | -8.2272 (11.6158)
  Day 85 - Spot 2: number analyzed (Participants) | 17
  Day 85 - Spot 2 | -7.6171 (16.1511)
  Day 85 - Spot 3: number analyzed (Participants) | 18
  Day 85 - Spot 3 | -13.1811 (14.4647)
  Day 113 - Spot 1: number analyzed (Participants) | 17
  Day 113 - Spot 1 | -8.0665 (11.9970)
  Day 113 - Spot 2: number analyzed (Participants) | 16
  Day 113 - Spot 2 | -9.2906 (13.7202)
  Day 113 - Spot 3: number analyzed (Participants) | 17
  Day 113 - Spot 3 | -11.2776 (12.9322)
  Day 155 - Spot 1: number analyzed (Participants) | 14
  Day 155 - Spot 1 | -7.0229 (15.4066)
  Day 155 - Spot 2: number analyzed (Participants) | 13
  Day 155 - Spot 2 | -7.0408 (12.8562)
  Day 155 - Spot 3: number analyzed (Participants) | 14
  Day 155 - Spot 3 | -10.4414 (14.5146)
  Day 197 - Spot 1: number analyzed (Participants) | 16
  Day 197 - Spot 1 | -8.9200 (11.3266)
  Day 197 - Spot 2: number analyzed (Participants) | 15
  Day 197 - Spot 2 | -11.2953 (15.3452)
  Day 197 - Spot 3: number analyzed (Participants) | 16
  Day 197 - Spot 3 | -11.1625 (16.2087)

28. Secondary Outcome: Percent Change From Baseline in TEWL Before STS on Normal Skin in Healthy Volunteers at Days 8, 15, 22, 29, 43, 57, 85, 113, 155 and 197
Description: TEWL assessment: noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. Normal skin areas for TEWL assessment were identified at baseline (predefined skin area). Within predefined normal skin areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS on pre-defined normal skin areas at specified time points. At each visit, before STS, all three spots were assessed. Percent change from Baseline at specified time points in TEWL before STS on normal skin (at each spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Days 8, 15, 22, 29, 43, 57, 85, 113, 155 and 197
Population: Analysis was performed on mITT population. Here, 'number analyzed' = participants with available data for each specified category. Data for this OM was not planned to be collected and analyzed for 'atopic dermatitis participant' arm as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 15
percent change
  Day 8 - Spot 1: number analyzed (Participants) | 13
  Day 8 - Spot 1 | 5.0103 (39.4170)
  Day 8 - Spot 2: number analyzed (Participants) | 13
  Day 8 - Spot 2 | -8.7688 (20.5764)
  Day 8 - Spot 3: number analyzed (Participants) | 13
  Day 8 - Spot 3 | -3.8203 (19.5160)
  Day 15 - Spot 1: number analyzed (Participants) | 14
  Day 15 - Spot 1 | 1.9837 (27.7012)
  Day 15 - Spot 2: number analyzed (Participants) | 14
  Day 15 - Spot 2 | -4.0758 (22.1886)
  Day 15 - Spot 3: number analyzed (Participants) | 14
  Day 15 - Spot 3 | -1.7489 (21.1652)
  Day 22 - Spot 1: number analyzed (Participants) | 12
  Day 22 - Spot 1 | -2.6655 (19.8558)
  Day 22 - Spot 2: number analyzed (Participants) | 12
  Day 22 - Spot 2 | 7.5939 (22.7859)
  Day 22 - Spot 3: number analyzed (Participants) | 12
  Day 22 - Spot 3 | 3.8603 (12.1068)
  Day 29 - Spot 1: number analyzed (Participants) | 13
  Day 29 - Spot 1 | -1.7648 (21.4820)
  Day 29 - Spot 2: number analyzed (Participants) | 13
  Day 29 - Spot 2 | 9.9969 (14.4219)
  Day 29 - Spot 3: number analyzed (Participants) | 13
  Day 29 - Spot 3 | 8.4098 (15.2499)
  Day 43 - Spot 1: number analyzed (Participants) | 14
  Day 43 - Spot 1 | 1.4115 (27.8012)
  Day 43 - Spot 2: number analyzed (Participants) | 14
  Day 43 - Spot 2 | 2.9668 (30.1272)
  Day 43 - Spot 3: number analyzed (Participants) | 14
  Day 43 - Spot 3 | 13.4093 (35.9985)
  Day 57 - Spot 1: number analyzed (Participants) | 12
  Day 57 - Spot 1 | 7.6533 (24.0747)
  Day 57 - Spot 2: number analyzed (Participants) | 12
  Day 57 - Spot 2 | 5.3384 (17.9065)
  Day 57 - Spot 3: number analyzed (Participants) | 12
  Day 57 - Spot 3 | 12.6926 (24.7125)
  Day 85 - Spot 1: number analyzed (Participants) | 14
  Day 85 - Spot 1 | 5.2021 (23.1397)
  Day 85 - Spot 2: number analyzed (Participants) | 14
  Day 85 - Spot 2 | 0.7096 (19.5448)
  Day 85 - Spot 3: number analyzed (Participants) | 14
  Day 85 - Spot 3 | 5.1021 (20.0690)
  Day 113 - Spot 1: number analyzed (Participants) | 11
  Day 113 - Spot 1 | 2.6054 (26.2241)
  Day 113 - Spot 2: number analyzed (Participants) | 11
  Day 113 - Spot 2 | 9.4234 (24.1533)
  Day 113 - Spot 3: number analyzed (Participants) | 11
  Day 113 - Spot 3 | 17.0905 (16.4596)
  Day 155 - Spot 1 | 10.3105 (52.8138)
  Day 155 - Spot 2 | 11.2398 (22.7028)
  Day 155 - Spot 3 | 11.5842 (27.2298)
  Day 197 - Spot 1 | 3.3636 (26.9400)
  Day 197 - Spot 2 | 5.3772 (19.9583)
  Day 197 - Spot 3 | 12.0900 (24.8690)

29. Secondary Outcome: Absolute Change From Baseline in TEWL Before STS on Normal Skin in Healthy Volunteers at Days 8, 15, 22, 29, 43, 57, 85, 113, 155 and 197
Description: TEWL assessment: noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. Normal skin areas for TEWL assessment were identified at baseline (predefined skin area). Within predefined normal skin areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS on pre-defined normal skin areas at specified time points. At each visit, before STS, all three spots were assessed. Absolute change from baseline at specified time points in TEWL before STS on normal skin (at each spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Days 8, 15, 22, 29, 43, 57, 85, 113, 155 and 197
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 15
grams per square meter per hour
  Day 8 - Spot 1: number analyzed (Participants) | 13
  Day 8 - Spot 1 | -0.2508 (4.8798)
  Day 8 - Spot 2: number analyzed (Participants) | 13
  Day 8 - Spot 2 | -1.8215 (3.3907)
  Day 8 - Spot 3: number analyzed (Participants) | 13
  Day 8 - Spot 3 | -0.7869 (2.9791)
  Day 15 - Spot 1: number analyzed (Participants) | 14
  Day 15 - Spot 1 | -0.5786 (3.3947)
  Day 15 - Spot 2: number analyzed (Participants) | 14
  Day 15 - Spot 2 | -1.0029 (3.4320)
  Day 15 - Spot 3: number analyzed (Participants) | 14
  Day 15 - Spot 3 | -0.3829 (3.3925)
  Day 22 - Spot 1: number analyzed (Participants) | 12
  Day 22 - Spot 1 | -0.7575 (3.2991)
  Day 22 - Spot 2: number analyzed (Participants) | 12
  Day 22 - Spot 2 | 1.0233 (3.7207)
  Day 22 - Spot 3: number analyzed (Participants) | 12
  Day 22 - Spot 3 | 0.6433 (2.0759)
  Day 29 - Spot 1: number analyzed (Participants) | 13
  Day 29 - Spot 1 | -1.1631 (3.1429)
  Day 29 - Spot 2: number analyzed (Participants) | 13
  Day 29 - Spot 2 | 0.8585 (1.8609)
  Day 29 - Spot 3: number analyzed (Participants) | 13
  Day 29 - Spot 3 | 0.7938 (1.7624)
  Day 43 - Spot 1: number analyzed (Participants) | 14
  Day 43 - Spot 1 | -1.0129 (4.0940)
  Day 43 - Spot 2: number analyzed (Participants) | 14
  Day 43 - Spot 2 | -0.8357 (4.7103)
  Day 43 - Spot 3: number analyzed (Participants) | 14
  Day 43 - Spot 3 | 0.7057 (5.1247)
  Day 57 - Spot 1: number analyzed (Participants) | 12
  Day 57 - Spot 1 | 0.6308 (4.1304)
  Day 57 - Spot 2: number analyzed (Participants) | 12
  Day 57 - Spot 2 | 0.2283 (2.6839)
  Day 57 - Spot 3: number analyzed (Participants) | 12
  Day 57 - Spot 3 | 1.5142 (4.1943)
  Day 85 - Spot 1: number analyzed (Participants) | 14
  Day 85 - Spot 1 | 0.0164 (3.2348)
  Day 85 - Spot 2: number analyzed (Participants) | 14
  Day 85 - Spot 2 | -0.3221 (3.5460)
  Day 85 - Spot 3: number analyzed (Participants) | 14
  Day 85 - Spot 3 | 0.2779 (3.8491)
  Day 113 - Spot 1: number analyzed (Participants) | 11
  Day 113 - Spot 1 | -0.3791 (3.4231)
  Day 113 - Spot 2: number analyzed (Participants) | 11
  Day 113 - Spot 2 | 0.4882 (2.5528)
  Day 113 - Spot 3: number analyzed (Participants) | 11
  Day 113 - Spot 3 | 2.0527 (2.1762)
  Day 155 - Spot 1 | -0.9293 (6.5972)
  Day 155 - Spot 2 | 0.6880 (3.7653)
  Day 155 - Spot 3 | 0.4793 (4.5057)
  Day 197 - Spot 1 | -0.6153 (4.8187)
  Day 197 - Spot 2 | -0.0427 (3.6560)
  Day 197 - Spot 3 | 0.6747 (4.8536)

30. Secondary Outcome: Percent Change From Baseline in Area Under the Curve (AUC) of TEWL on Lesional Skin in AD Participants at Days 57, 113 and 197
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. TEWL AUC done over defined number of STS was used to reflect the overall integrity of the stratum corneum. LS areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within the predefined LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS areas at specified time points. TEWL AUC was a composite measure before and after 5, 10, 15 and 20 STS at each specified time point. AUC of TEWL: calculated for each visit using trapezoidal method. STS assessment at baseline (Week 0, Day 1), Days 57, 113 and 197 was conducted on first spot. Percent change from baseline at specified time points in TEWL AUC (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Days 57, 113 and 197
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' = participants with available data for this OM and 'number analyzed' = participants with available data for each specified category. Data for this OM was not planned to be collected and analyzed for 'healthy volunteer' arm as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 19
percent change
  Day 57 | -38.2091 (25.6654)
  Day 113: number analyzed (Participants) | 18
  Day 113 | -34.0025 (29.1866)
  Day 197: number analyzed (Participants) | 15
  Day 197 | -40.0143 (26.9737)

31. Secondary Outcome: Absolute Change From Baseline in AUC of TEWL on Lesional Skin in AD Participants at Days 57, 113 and 197
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum to characterize SBF. TEWL combined with STS measures SBF. TEWL AUC done over defined number of STS (nsts) used to reflect the overall integrity of stratum corneum. LS areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within predefined LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS areas at specified time points. TEWL AUC was a composite measure before and after 5, 10, 15 and 20 STS at each specified time point. AUC of TEWL: calculated for each visit using trapezoidal method. STS assessment at baseline (Week 0, Day 1), Days 57, 113 and 197 was conducted on first spot. Absolute change from baseline at specified time points in TEWL AUC (first spot) in AD participants reported in this OM.
Time Frame: Baseline, Days 57, 113 and 197
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: nsts*grams per square meter per hour
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 19
nsts*grams per square meter per hour
  Day 57 | -632.0224 (494.4981)
  Day 113: number analyzed (Participants) | 18
  Day 113 | -608.1875 (601.7999)
  Day 197: number analyzed (Participants) | 15
  Day 197 | -659.4033 (570.2425)

32. Secondary Outcome: Percent Change From Baseline in AUC of TEWL on Non-lesional Skin in AD Participants at Days 57, 113 and 197
Description: TEWL assessment: noninvasive in vivo measurement of water loss across stratum corneum used to characterize SBF. TEWL combined with STS measures SBF. TEWL AUC done over defined number of STS reflect the overall integrity of the stratum corneum. Non-LS areas for TEWL assessment & STS were identified at baseline (predefined skin area). Within predefined non-LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL measured prior to STS & after 5, 10, 15 & 20 STS on pre-defined non-LS areas at specified time points. TEWL AUC was a composite measure before & after 5, 10, 15 &20 STS at each specified time point. AUC of TEWL: calculated for each visit using trapezoidal method. STS assessment at baseline (Week 0, Day 1), Days 57, 113 & 197 was conducted on first spot. Percent change from baseline at specified time points in TEWL AUC (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Days 57, 113 and 197
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 19
percent change
  Day 57 | -21.7570 (29.1137)
  Day 113: number analyzed (Participants) | 17
  Day 113 | -10.8940 (50.7679)
  Day 197: number analyzed (Participants) | 16
  Day 197 | -28.6897 (26.0253)

33. Secondary Outcome: Absolute Change From Baseline in AUC of TEWL on Non-lesional Skin in AD Participants at Days 57, 113 and 197
Description: TEWL assessment: a noninvasive in vivo measurement of water loss across stratum corneum to characterize SBF. TEWL combined with STS measures SBF. TEWL AUC done over defined number of STS used to reflect the overall integrity of stratum corneum. Non-LS areas for TEWL assessment and STS were identified at baseline(predefined skin area). Within predefined non-LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10,15 and 20 STS on pre-defined non-LS areas at specified time points. TEWL AUC was a composite measure before and after 5, 10, 15 and 20 STS at each specified time point. AUC of TEWL: calculated for each visit using trapezoidal method. STS assessment at baseline(Week 0, Day 1), Days 57, 113 and 197 was conducted on first spot. Absolute change from baseline at specified time points in TEWL AUC (first spot) in AD participants reported in this OM.
Time Frame: Baseline, Days 57, 113 and 197
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: nsts*grams per square meter per hour
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 19
nsts*grams per square meter per hour
  Day 57 | -281.9579 (342.1271)
  Day 113: number analyzed (Participants) | 17
  Day 113 | -217.7544 (462.0173)
  Day 197: number analyzed (Participants) | 16
  Day 197 | -367.5469 (340.1948)

34. Secondary Outcome: Percent Change From Baseline in AUC of TEWL on Normal Skin in Healthy Volunteers at Days 57, 113 and 197
Description: TEWL: noninvasive in vivo measurement of water loss across stratum corneum to characterize SBF. TEWL combined with STS measures SBF. TEWL AUC done over a defined number of STS used to reflect the overall integrity of the stratum corneum. Normal skin areas for TEWL assessment & STS were identified at baseline(predefined skin area). Within predefined normal skin areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL measured prior to STS & after 5, 10,15 & 20 STS on pre-defined normal skin areas at specified time points. TEWL AUC: composite measure before & after 5, 10, 15& 20 STS at each specified time point. AUC of TEWL: calculated for each visit using trapezoidal method. STS assessment at baseline (Week 0, Day 1), Days 57, 113 & 197 conducted on first spot. Percent Change from baseline at specified time points in TEWL AUC (first spot) in healthy volunteers reported in this OM.
Time Frame: Baseline, Days 57, 113 and 197
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' = participants with available data for this OM and 'number analyzed' = participants with available data for each specified category. Data for this OM was not planned to be collected and analyzed for 'atopic dermatitis participant' arm as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 15
percent change
  Day 57: number analyzed (Participants) | 12
  Day 57 | 3.2794 (15.6493)
  Day 113: number analyzed (Participants) | 11
  Day 113 | 3.4753 (30.2504)
  Day 197 | -10.1582 (18.4753)

35. Secondary Outcome: Absolute Change From Baseline in AUC of TEWL on Normal Skin in Healthy Volunteers at Days 57, 113 and 197
Description: TEWL: noninvasive in vivo measurement of water loss across stratum corneum to characterize SBF. TEWL combined with STS measures SBF. TEWL AUC done over defined number of STS used to reflect the overall integrity of stratum corneum. Normal skin areas for TEWL assessment and STS identified at baseline(predefined skin area). Within predefined Normal skin areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL measured prior to STS and after 5, 10,15 and 20 STS on pre-defined Normal skin areas at specified time points. TEWL AUC was a composite measure before and after 5, 10,15 and 20 STS at each specified time point. AUC of TEWL: calculated for each visit using trapezoidal method. STS assessment at baseline (Week 0, Day 1), Days 57, 113 and 197 conducted on first spot. Percent change from baseline at specified time points in TEWL AUC (first spot) in healthy volunteers reported in this OM.
Time Frame: Baseline, Days 57, 113 and 197
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: nsts*grams per square meter per hour
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 15
nsts*grams per square meter per hour
  Day 57: number analyzed (Participants) | 12
  Day 57 | 16.8563 (70.4582)
  Day 113: number analyzed (Participants) | 11
  Day 113 | 2.5568 (197.8379)
  Day 197 | -72.9050 (108.8230)

36. Secondary Outcome: Percent Change From Baseline in TEWL After 5, 10, 15 and 20 STS on Lesional Skin in AD Participants at Days 57, 113 and 197
Description: TEWL assessment: noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of skin are peeled away using adhesive discs. LS areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within predefined LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL: measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS areas at specified time points. STS assessment at baseline (Week 0, Day 1), Day 57, 113 and 197 were conducted on first spot. Percent change from baseline at specified time points in TEWL after STS on LS (first spot) in AD participant were reported in this OM.
Time Frame: Baseline, Days 57, 113 and 197
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 19
percent change
  After 5 STS: Day 57 | -42.2019 (22.5314)
  After 5 STS: Day 113: number analyzed (Participants) | 18
  After 5 STS: Day 113 | -38.5633 (27.1211)
  After 5 STS: Day 197: number analyzed (Participants) | 15
  After 5 STS: Day 197 | -36.4601 (47.5902)
  After 10 STS: Day 57: number analyzed (Participants) | 18
  After 10 STS: Day 57 | -40.4595 (27.4572)
  After 10 STS: Day 113: number analyzed (Participants) | 17
  After 10 STS: Day 113 | -34.7741 (31.0541)
  After 10 STS: Day 197: number analyzed (Participants) | 13
  After 10 STS: Day 197 | -39.9440 (29.2084)
  After 15 STS: Day 57 | -41.6561 (24.0960)
  After 15 STS: Day 113: number analyzed (Participants) | 18
  After 15 STS: Day 113 | -33.3119 (32.7125)
  After 15 STS: Day 197: number analyzed (Participants) | 14
  After 15 STS: Day 197 | -38.4286 (27.0978)
  After 20 STS: Day 57 | -34.8297 (23.0520)
  After 20 STS: Day 113: number analyzed (Participants) | 17
  After 20 STS: Day 113 | -33.1336 (28.1613)
  After 20 STS: Day 197: number analyzed (Participants) | 14
  After 20 STS: Day 197 | -35.6561 (23.0987)

37. Secondary Outcome: Absolute Change From Baseline in TEWL After 5, 10, 15 and 20 STS on Lesional Skin in AD Participants at Days 57, 113 and 197
Description: TEWL assessment: noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, the uppermost layers of skin are peeled away using adhesive discs. LS areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within predefined LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL: measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined LS areas at specified time points. STS assessment at baseline (Week 0, Day 1), Day 57, 113 and 197 was conducted on first spot. Absolute change from baseline at specified time points in TEWL after STS on LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Days 57, 113 and 197
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 19
grams per square meter per hour
  After 5 STS: Day 57 | -31.3795 (25.4943)
  After 5 STS: Day 113: number analyzed (Participants) | 18
  After 5 STS: Day 113 | -31.1761 (31.3420)
  After 5 STS: Day 197: number analyzed (Participants) | 15
  After 5 STS: Day 197 | -33.5753 (40.1857)
  After 10 STS: Day 57: number analyzed (Participants) | 18
  After 10 STS: Day 57 | -36.4267 (31.1758)
  After 10 STS: Day 113: number analyzed (Participants) | 17
  After 10 STS: Day 113 | -33.1024 (36.2286)
  After 10 STS: Day 197: number analyzed (Participants) | 13
  After 10 STS: Day 197 | -35.8254 (33.3362)
  After 15 STS: Day 57 | -37.9779 (23.3049)
  After 15 STS: Day 113: number analyzed (Participants) | 18
  After 15 STS: Day 113 | -33.4028 (31.1957)
  After 15 STS: Day 197: number analyzed (Participants) | 14
  After 15 STS: Day 197 | -36.0843 (27.5612)
  After 20 STS: Day 57 | -35.0726 (23.5765)
  After 20 STS: Day 113: number analyzed (Participants) | 17
  After 20 STS: Day 113 | -35.6671 (31.2267)
  After 20 STS: Day 197: number analyzed (Participants) | 14
  After 20 STS: Day 197 | -34.5257 (23.9001)

38. Secondary Outcome: Percent Change From Baseline in TEWL After 5, 10, 15 and 20 STS on Non-lesional Skin in AD Participants at Days 57, 113 and 197
Description: TEWL assessment: noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, uppermost layers of skin are peeled away using adhesive discs. Non-LS areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within predefined non-LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL: measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined non-LS areas at specified time points. STS assessment at baseline (Week 0, Day 1), Day 57, 113and 197 was conducted on first spot. Percent change from baseline at specified time points in TEWL after STS on non-LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Days 57, 113 and 197
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 19
percent change
  After 5 STS: Day 57 | -24.8218 (31.4633)
  After 5 STS: Day 113: number analyzed (Participants) | 17
  After 5 STS: Day 113 | -4.8842 (70.5670)
  After 5 STS: Day 197: number analyzed (Participants) | 16
  After 5 STS: Day 197 | -29.7635 (44.0691)
  After 10 STS: Day 57 | -20.3640 (43.5318)
  After 10 STS: Day 113: number analyzed (Participants) | 17
  After 10 STS: Day 113 | -3.8193 (74.6263)
  After 10 STS: Day 197: number analyzed (Participants) | 16
  After 10 STS: Day 197 | -29.6888 (38.9536)
  After 15 STS: Day 57 | -18.4348 (33.3647)
  After 15 STS: Day 113: number analyzed (Participants) | 17
  After 15 STS: Day 113 | -7.6067 (54.7945)
  After 15 STS: Day 197: number analyzed (Participants) | 16
  After 15 STS: Day 197 | -27.2268 (25.1580)
  After 20 STS: Day 57 | -19.2584 (30.1343)
  After 20 STS: Day 113: number analyzed (Participants) | 17
  After 20 STS: Day 113 | -6.1452 (67.9496)
  After 20 STS: Day 197: number analyzed (Participants) | 16
  After 20 STS: Day 197 | -22.3311 (23.0908)

39. Secondary Outcome: Secondary: Absolute Change From Baseline in TEWL After 5, 10, 15 and 20 STS on Non-lesional Skin in AD Participants at Days 57, 113 and 197
Description: TEWL assessment: noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, uppermost layers of skin are peeled away using adhesive discs. Non-LS areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within predefined non-LS areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL: measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined non-LS areas at specified time points. STS assessment at baseline (Week 0, Day 1), Day 57, 113 and 197 was conducted on the first spot. Absolute change from baseline at specified time points in TEWL after STS on non-LS (first spot) in AD participants were reported in this OM.
Time Frame: Baseline, Days 57, 113 and 197
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Atopic Dermatitis Participants
Number analyzed (Participants) | 19
grams per square meter per hour
  After 5 STS: Day 57 | -11.8526 (12.6180)
  After 5 STS: Day 113: number analyzed (Participants) | 17
  After 5 STS: Day 113 | -9.0771 (21.3022)
  After 5 STS: Day 197: number analyzed (Participants) | 16
  After 5 STS: Day 197 | -15.8375 (18.0369)
  After 10 STS: Day 57 | -15.0005 (20.1721)
  After 10 STS: Day 113: number analyzed (Participants) | 17
  After 10 STS: Day 113 | -10.9488 (31.1300)
  After 10 STS: Day 197: number analyzed (Participants) | 16
  After 10 STS: Day 197 | -21.2825 (23.2998)
  After 15 STS: Day 57 | -16.1047 (26.4807)
  After 15 STS: Day 113: number analyzed (Participants) | 17
  After 15 STS: Day 113 | -12.6576 (30.0412)
  After 15 STS: Day 197: number analyzed (Participants) | 16
  After 15 STS: Day 197 | -21.9006 (19.2885)
  After 20 STS: Day 57 | -18.5800 (30.3574)
  After 20 STS: Day 113: number analyzed (Participants) | 17
  After 20 STS: Day 113 | -13.6682 (33.3065)
  After 20 STS: Day 197: number analyzed (Participants) | 16
  After 20 STS: Day 197 | -20.0575 (16.1537)

40. Secondary Outcome: Percent Change From Baseline in TEWL After 5, 10, 15 and 20 STS on Normal Skin in Healthy Volunteers at Days 57, 113 and 197
Description: TEWL assessment: noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, uppermost layers of skin are peeled away using adhesive discs. Normal skin areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within predefined normal skin areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment at baseline (Week 0, Day 1), Day 57, 113 and 197 was conducted on first spot. Percent change from baseline at specified time points in TEWL after STS on normal skin (first spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Days 57, 113 and 197
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 15
percent change
  After 5 STS: Day 57: number analyzed (Participants) | 12
  After 5 STS: Day 57 | 4.9595 (16.0950)
  After 5 STS: Day 113: number analyzed (Participants) | 11
  After 5 STS: Day 113 | 1.4464 (26.7257)
  After 5 STS: Day 197 | -1.6729 (25.2293)
  After 10 STS: Day 57: number analyzed (Participants) | 12
  After 10 STS: Day 57 | 4.0996 (20.4647)
  After 10 STS: Day 113: number analyzed (Participants) | 11
  After 10 STS: Day 113 | 0.7091 (25.0615)
  After 10 STS: Day 197 | -7.4475 (19.7215)
  After 15 STS: Day 57: number analyzed (Participants) | 12
  After 15 STS: Day 57 | 3.2339 (20.9086)
  After 15 STS: Day 113: number analyzed (Participants) | 11
  After 15 STS: Day 113 | 4.5364 (42.7525)
  After 15 STS: Day 197 | -14.0103 (18.5552)
  After 20 STS: Day 57: number analyzed (Participants) | 12
  After 20 STS: Day 57 | 4.3494 (27.5527)
  After 20 STS: Day 113: number analyzed (Participants) | 11
  After 20 STS: Day 113 | 13.2578 (64.3880)
  After 20 STS: Day 197 | -18.0480 (22.6193)

41. Secondary Outcome: Absolute Change From Baseline in TEWL After 5, 10, 15 and 20 STS on Normal Skin in Healthy Volunteers at Days 57, 113 and 197
Description: TEWL assessment: noninvasive in vivo measurement of water loss across stratum corneum that is used to characterize SBF. TEWL combined with STS measures SBF. With STS, uppermost layers of skin are peeled away using adhesive discs. Normal skin areas for TEWL assessment and STS were identified at baseline (predefined skin area). Within predefined normal skin areas, 3 closely adjacent non-overlapping spots were identified for subsequent SBF assessment. TEWL was measured prior to STS and after 5, 10, 15 and 20 STS on pre-defined normal skin areas at specified time points. STS assessment at baseline (Week 0, Day 1), Day 57, 113 and 197 were conducted on first spot. Absolute change from baseline at specified time points in TEWL after STS on normal skin (first spot) in healthy volunteers were reported in this OM.
Time Frame: Baseline, Days 57, 113 and 197
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: grams per square meter per hour
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 15
grams per square meter per hour
  After 5 STS: Day 57: number analyzed (Participants) | 12
  After 5 STS: Day 57 | 0.5642 (3.3355)
  After 5 STS: Day 113: number analyzed (Participants) | 11
  After 5 STS: Day 113 | -1.0255 (4.3657)
  After 5 STS: Day 197 | -1.5627 (5.2934)
  After 10 STS: Day 57: number analyzed (Participants) | 12
  After 10 STS: Day 57 | 0.2825 (4.5142)
  After 10 STS: Day 113: number analyzed (Participants) | 11
  After 10 STS: Day 113 | -1.3482 (6.6778)
  After 10 STS: Day 197 | -3.0880 (5.2754)
  After 15 STS: Day 57: number analyzed (Participants) | 12
  After 15 STS: Day 57 | 0.4750 (6.4442)
  After 15 STS: Day 113: number analyzed (Participants) | 11
  After 15 STS: Day 113 | 0.1082 (17.5865)
  After 15 STS: Day 197 | -5.8847 (8.1968)
  After 20 STS: Day 57: number analyzed (Participants) | 12
  After 20 STS: Day 57 | 3.4683 (9.8235)
  After 20 STS: Day 113: number analyzed (Participants) | 11
  After 20 STS: Day 113 | 5.9327 (32.0123)
  After 20 STS: Day 197 | -7.4760 (9.3514)

ADVERSE EVENTS:
Time Frame: For AD participants: from first dose (i.e., Day 1) of IMP administration up to end of treatment visit (i.e., Day 113). For healthy volunteers: from signature of consent form to end of study (i.e., up to Day 197)
Description: Analysis was performed on safety population that included all participants, who actually received at least 1 dose of IMP or had at least 1 TEWL/STS assessment and all healthy volunteers who have at least 1 TEWL/STS assessment performed.
Groups:
- Atopic Dermatitis Participant: Pediatric participants with moderate-to-severe AD and with baseline body weight >=15 kg and <30 kg received a SC loading dose of dupilumab 600 mg (2 injections of dupilumab 300 mg) on Day 1 (Week 0) followed by dupilumab 300 mg SC injection Q4W, from Week 4 to Week 12. Pediatric participants with body weight >=30 kg and <60 kg received SC loading dose of dupilumab 400 mg (2 injections of dupilumab 200 mg) on Day 1 (Week 0), followed by dupilumab 200 mg SC injection Q2W, from Week 2 to Week 14.
Arm/Group | Healthy Volunteers | Atopic Dermatitis Participant
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/23
Other Adverse Events (participants affected / at risk) | 6/18 | 21/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers (N=18) | Atopic Dermatitis Participant (N=23)
Covid-19 (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Dermatitis Infected (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal Viral Infection (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Molluscum Contagiosum (Infections and infestations) | 0 (0) | 1 (1)
Otitis Media Chronic (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Skin Bacterial Infection (Infections and infestations) | 1 (1) | 0 (0)
Suspected Covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 4 (5)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Food Allergy (Immune system disorders) | 0 (0) | 1 (1)
Seasonal Allergy (Immune system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (4)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 0 (0) | 1 (1)
Eye Irritation (Eye disorders) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 0 (0) | 1 (1)
Eye Pruritus (Eye disorders) | 0 (0) | 2 (2)
Ocular Hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Vision Blurred (Eye disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (10)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Medical Device Site Haemorrhage (General disorders) | 0 (0) | 6 (7)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Arthropod Sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT04718870/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT04718870/SAP_001.pdf